CLINICAL TRIAL: NCT00430742
Title: A Phase III Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Efficacy of Taranabant (MK0364) in Overweight and Obese Patients With Type 2 Diabetes Mellitus (T2DM) Followed by a 1-Year Extension
Brief Title: An Investigational Drug Study to Assess Weight Loss in Patients With Type 2 Diabetes Mellitus (0364-011)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The overall profile does not support development for obesity
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0364-011; 2006_021
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Obesity Type 2 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Arm 1: MK0364 0.5 mg capsule once daily
  Interventions: Drug: Taranabant
- 2 (Experimental): Arm 2: MK0364 1 mg capsule once daily
  Interventions: Drug: Taranabant
- 3 (Experimental): Arm 3: MK0364 2 mg capsule once daily
  Interventions: Drug: Taranabant
- 4 (Placebo Comparator): Arm 4: Pbo capsule once daily
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Taranabant — Taranabant 0.5 mg, 1 mg capsule, 2 mg capsule once daily Treatment for 52 weeks.
  Arms: 1; 2; 3
Drug: Comparator: Placebo — Placebo capsule once daily. Treatment for 52 weeks.
  Arms: 4

SUMMARY:
A worldwide study with extension in patients with type 2 diabetes mellitus to assess the safety and tolerability as well as the effects of treatment with an investigational drug for weight loss on body weight.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 27 kg/m2 and 43 kg/m2 and HbA1c between 7.0% and 10%

Exclusion Criteria:

* History of major psychiatric disorder
* Blood pressure greater than 160/100
* Use of any antihyperglycemic agent other than metformin
* Triglycerides greater then 600 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Body weight at 36 weeks, HbA1c at 36 weeks | 36 weeks

SECONDARY OUTCOMES:
Body weight at 24 and 52 weeks, HbA1c at 24 and 52 weeks | 24 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Kipnes MS, Hollander P, Fujioka K, Gantz I, Seck T, Erondu N, Shentu Y, Lu K, Suryawanshi S, Chou M, Johnson-Levonas AO, Heymsfield SB, Shapiro D, Kaufman KD, Amatruda JM. A one-year study to assess the safety and efficacy of the CB1R inverse agonist taranabant in overweight and obese patients with type 2 diabetes. Diabetes Obes Metab. 2010 Jun;12(6):517-31. doi: 10.1111/j.1463-1326.2009.01188.x. PMID 20518807